CLINICAL TRIAL: NCT02141802
Title: Clinical Effectiveness of Increased Standing Time in Non-ambulant Children With Cerebral Palsy:a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rachel Rapson (Other)
Collaborators: University of Plymouth (Other)
Responsible Party: Sponsor-Investigator, Rachel Rapson, Research Assistant, University of Plymouth
Organization: University of Plymouth (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC 13/SW/0228
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Cerebral Palsy; Developmental Delay
MeSH Terms: conditions — Cerebral Palsy; Learning Disabilities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Normal standing time
  Interventions: Behavioral: control
- Doubling standing time (Experimental): Doubled standing time calculated by doubling baseline standing time
  Interventions: Behavioral: Doubling standing time

INTERVENTIONS:
Behavioral: Doubling standing time — Doubling standing time using child's previously prescribed standing frame with a progression of 10% increase in time/month up to 2 hrs/day maximum
  Arms: Doubling standing time
Behavioral: control — Continue with usual standing time with a progression of 10% increase in time/month up to 1 hr/day maximum
  Arms: Control

SUMMARY:
Children with cerebral palsy commonly use standing frames to position them to help prevent contracture and deformity and to help their function. There is a lack of evidence to support the correct dosage of standing frame use.

The aim of this study is to pilot a randomised controlled trial of the clinical effects of doubling the duration of standing, using standing frames, in young children who are unable to walk, who have cerebral palsy or developmental delay.

It will determine whether it is feasable to carry out a multi-centred trial.

The study objectives will be to determine:

1. presence of adverse events
2. recruitment and drop out rate
3. compliance with the intervention
4. feasibility of the randomisation and minimisation process
5. the proportion of the outcome measures taken
6. effect size estimate
7. required study costs
8. effectiveness of blinding procedure

DETAILED DESCRIPTION:
Thirty non-ambulant children with cerebral palsy will be randomised into one of two groups that either (a) maintains the child's current standing frame program- the control group (n=15) (b) doubles the standing time- the intervention group (n=15). Outcome measures will be taken at baseline and at 6 monthly intervals by a blinded assessor.

Research process and flow Families who are willing to participate in the study will be provided with a diary sheet that will allow them to record over a baseline 2 week period how frequently their child stood and in what position. The diary sheet will be available in word or hard copy format. An e mail/ stamped addressed envelope will be provided to return the diary at the end of 2 weeks. Participants will be reminded via text/ phone / e mail (depending on their preferred method of communication) after 1 week if they have not returned their diary sheets.

On receipt of the diary sheets participants will be randomized into an intervention or control group (see below). A therapist will explain the group allocation to the families at their home or their local CDC. The trial will run for 12 months with the outcome measures being taken by an assessor blinded to group allocation. The primary outcome measure (hip migration percentage) will be taken at 0 and 12 months so as to fit in with practice across the South West and not to increase x ray exposure. The secondary outcome measures will be taken at baseline, 6 and 12 months. The final RCT will involve a 3 yr follow-up phase.

Sample Size We aim to recruit 15 people per group. An audit of CDC records suggests that there are between 5-6 eligible participants over a 12 month recruitment period. With 8 main recruitment centres this would result in 40-48 potential participants and a required recruitment rate of 75-63%. An on-going study looking at walking in children with older children with CP at Plymouth University suggests that this recruitment rate is feasible. Determining the actual recruitment rate in this particular patient population and the feasibility of using multiple centres across one region is one objective of the pilot study.

Randomisation

Thirty children with Cerebral Palsy (age 1-12 yrs; GMFCS III-V) will be recruited from South West based services. Participants will be randomly allocated to the intervention or control using a web-based system. A minimisation algorithm will be used to ensure balance between the groups on the basis of the following:

* Age (<6 yrs Vs >6 yrs)
* Functional ability (GMFCS=III or IVs GMFCS =V)
* Baseline standing time (<30 mins Vs >30 mins)

Intervention All participants will already be performing a standing regime as prescribed by their treating therapist. The study design and group allocation will be explained by the research assistant (RA1) either at the local CDC or at the participants' home. The control group will continue their usual standing-frame based regime. The intervention group will double their daily standing-frame time.

In both groups a guidance sheet will be provided about how to progress their standing time for the duration of the trial by 10%/month up to a maximum of 1 hr/day in the control group and 2 hr/day in the intervention group. Following PPI advice the guidance will be personalised to include photos of how to set their child up in their own standing frame and the correct position of supportive straps / correct posture to adopt.

The research assistant will visit both groups at the start of the trial and every 3 months. At each visit they will (a) check the position the child adopts in the standing frame (b) check footwear and splints for use and fit (c) check the progression of treatment (d) check and record any changes to their additional care routine by the treating therapist. Feedback about problems in footwear / splinting will be passed onto the child's treating therapist.

Outcome Measures The primary outcome measure will be taken at baseline (0 months) and at 12 months. This fits in with routine practice cross all centres in the South West although some centres take additional x-rays at 6 months. All other measures will be taken at 0, 6 and 12 months. Outcomes will be measured by an assessor blinded to the group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cerebral palsy or developmental delay
* Aged between 1-12 years at the beginning of the study
* Signs UMN involvement with spasticity or hypertonia in at least one limb
* Gross motor function classification III-V
* undertaking a standing programme of at least 1.5hours per week for at least a month

Exclusion Criteria:

* Soft tissue release that would require imobilization which would prevent standing within 6 months from the onset of the trial
* Bony surgery Soft that would require imobilization which would prevent standing within 12 months from the onset of the trial
* a fracture that would prevent standing

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Hip migration Percentage | baseline and 12 months
  In line with planned hip screening, not additional x rays.

SECONDARY OUTCOMES:
Standing time | weekly over 12 months
  By use of a daily diary
Muscle length | 0, 6 months and 12 months
  gastrocnemius, hamstrings and hip flexors
Rectus femoris circumference using ultrasound | 0, 6, 12 months
  1/3rd distance from proximal patella to ASIS. 3x cross section and 3 x longitudinal images taken and mean scores derived.
Muscle tone hip flexors hamstrings and ankle plantarflexors Tardieu test | 0, 6, 12 months
  3 range of movements at 100 degrees per second mean scores calculated
Muscle tone of gastrocnemius using the myotonometer | 0, 6, 12 months
  Muscle tap x 3 medial head of gastrocnemius at mid way between medial malleolus and head of the fibula. Mean score taken.
Paediatric pain profile | 0, 6 12 months
  parent reported structured score sheet
Gross motor function measure | 0, 6, 12 months
  standardised assessment GMFM66
CP CHILD questionnaire | 0, 6, 12 months
  parent reported questionairre

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Marsden, Phd, Principal Investigator — University of Plymouth
Locations (4):
- United Kingdom (4):
  - Royal Cornwall Hspitals Trust, Truro, Cornwall
  - Honeylands Specialist Child Assessment Centre, Exeter
  - Child Development centre, Plymouth Devon
  - John Parkes Unit Newton Road, Torbay